CLINICAL TRIAL: NCT06776809
Title: Effect of Music Listened During Toe Amputation on Patients' Anxiety, Pain, Sense of Safety and Surgical Fear
Brief Title: Effect of Music During Toe Amputation
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Afyonkarahisar Health Sciences University (Other)
Responsible Party: Principal Investigator, Yeliz Ciğerci, Assoc.Prof., Afyonkarahisar Health Sciences University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 2024/11
Record Dates: First submitted 2025-01-10; First posted 2025-01-15 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Amputation
Keywords: Amputation; Toe amputation; Music; Pain; Anxiety; Surgical fear; Sense of Safety
MeSH Terms: conditions — Pain; Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): Patients in the control group will not be allowed to listen to music. These patients will receive standard health care in the Diabetic Foot and Wound Care Clinic.
- Intervention Group- Listening to Sufi Music (Experimental): Patients in this group will listen to Sufi music during toe amputation in addition to standard health care in the Diabetic Foot and Wound Care Clinic. Music will be played to the patients with the help of Mp3 player and headphones throughout the operation. Disposable headphone covers will be used for the headphones and the covers will be changed for each patient.
  Interventions: Other: Music listening

INTERVENTIONS:
Other: Music listening — Selection of Sufi music will be played to the patients during the course of the operation.
  Arms: Intervention Group- Listening to Sufi Music

SUMMARY:
This randomized controlled intervention study aims to investigate the impact of music played during toe amputation on patients' anxiety, pain, sense of safety, and fear of surgery.

The study will be carried out with two groups: The control and the intervention groups with 60 participants for each group. While the control group participants will receive standard care, the intervention group participants will listen to selection of Sufi music during the whole amputation procedure in addition to standard care.

DETAILED DESCRIPTION:
Diabetes rates are continuing to rise worldwide, leading to an increasing number of people with diabetes seeking medical care for foot wounds, with approximately 35% of diabetic individuals experiencing a foot wound at some point in their lives. Diabetic foot (DF) wounds tend to recur, with a 50% recurrence rate after treatment. Foot wounds are responsible for 85% of amputations in diabetics, and the five-year mortality rate following a lower extremity amputation rises to 77%. It is estimated that a diabetic patient undergoes an amputation every 20 seconds globally. Lower extremity amputations encompass a range of procedures, from hemipelvectomy to toe amputations. Among the most common partial amputations are those of the big toe and other toes, with diabetes being the cause of about 24% of these amputations.

A comprehensive meta-analysis examined the risk factors for amputation associated with diabetic foot ulcers and found that the overall incidence of lower extremity amputation in diabetic foot ulcer patients is 31%. This study provides crucial epidemiological data for medical practice. Key risk factors associated with lower extremity amputation include male gender, smoking history, body mass index (BMI), hypertension, cardiovascular disease, kidney disease, white blood cell count, hemoglobin, and albumin levels. Among these factors, BMI, hemoglobin, and albumin levels were negatively correlated with the likelihood of amputation, while other factors, such as gender, smoking, and comorbidities, showed positive correlations.

These findings highlight the importance of monitoring and addressing these risk factors in patients with diabetic foot ulcers to reduce the likelihood of lower extremity amputations. Consequently, targeted preventive and intervention measures focusing on these risk factors are essential in clinical practice to improve patient outcomes.

The literature reveals that pain following lower extremity amputation is widespread and remains a significant factor affecting patients' quality of life. If not properly managed, this post-amputation pain can have detrimental consequences for the patient. Effective pain control during the perioperative period has been shown to help prevent chronic stump pain, highlighting the importance of intraoperative anesthesia management and postoperative acute pain control. These factors influence the body's stress response to surgery and have a direct impact on recovery, discharge, and the return to daily activities. This is particularly critical for amputation patients, as early mobilization plays a key role in both physical and psychological recovery.

These findings underscore the importance of managing perioperative pain in patients undergoing lower extremity amputation, especially during the early postoperative period. Uncontrolled postoperative pain is one of the primary risk factors for the development of chronic pain following surgery. For amputee patients, pain, particularly in the early stages after surgery, is often accompanied by significant emotional challenges. Therefore, for comprehensive care, it is essential to consider the interplay between pain experience and the emotional well-being of patients who have not received adequate pain management.The literature reveals that pain following lower extremity amputation is widespread and remains a significant factor affecting patients' quality of life. If not properly managed, this post-amputation pain can have detrimental consequences for the patient. Effective pain control during the perioperative period has been shown to help prevent chronic stump pain, highlighting the importance of intraoperative anesthesia management and postoperative acute pain control. These factors influence the body's stress response to surgery and have a direct impact on recovery, discharge, and the return to daily activities. This is particularly critical for amputation patients, as early mobilization plays a key role in both physical and psychological recovery.

These findings underscore the importance of managing perioperative pain in patients undergoing lower extremity amputation, especially during the early postoperative period. Uncontrolled postoperative pain is one of the primary risk factors for the development of chronic pain following surgery. For amputee patients, pain, particularly in the early stages after surgery, is often accompanied by significant emotional challenges. Therefore, for comprehensive care, it is essential to consider the interplay between pain experience and the emotional well-being of patients who have not received adequate pain management.

Anxiety often begins when an individual is informed that they require surgery and tends to increase during hospitalization. This heightened anxiety can negatively impact the individual's quality of life, their ability to adapt to the illness, and the overall progression of the condition. Surgical patients, in general, are considered to be at higher risk for experiencing anxiety.

A sense of safety is an inherent human need, and it is crucial for patients to feel safe within healthcare environments. While all healthcare practices aim to ensure patient safety, it is equally important to assess whether these practices foster a sense of safety for the patient. The sense of safety experienced by patients plays a vital role in their overall health and well-being.

To date, no studies have explored the effects of music on pain, anxiety, and the sense of safety in patients before, during, or after any type of amputation. Therefore, our study aims to investigate the impact of music played during toe amputation on patients' anxiety, pain, sense of safety, and fear of surgery.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or above,
* Having a toe amputation under spinal anesthesia due to diabetic foot,
* Without hearing/speech impairment,
* Without a diagnosis of psychiatric disorders,
* Without any professional training in music,
* and volunteered to participate.

Exclusion Criteria:

* Patients under 18 years of age,
* With hearing/speech impairment,
* With a diagnosis of psychiatric disorders,
* With any kind of professional training in music,
* and not willing to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-02-12 (Estimated); Primary Completion 2026-01-06 (Estimated); Study Completion 2026-01-06 (Estimated)

PRIMARY OUTCOMES:
Numerical Rating Scale-Anxiety (NRS-A) | 3 days
  The Numerical Rating Scale-Anxiety (NRS-A) has been widely used in research to assess anxiety levels, with its reliability and validity well-established. This scale, which ranges from 0 to 10, measures anxiety from "No Stress" (0) to "Very Bad Stress" (10). A higher score indicates a greater level of anxiety. The scale categorizes raw anxiety scores as follows: 0-no anxiety, 1-3-slightly anxious, 4-6-moderately anxious, 7-9-very or extremely anxious, and 10-the worst imaginable or extremely anxious.
Numerical Rating Scale-Pain (NRS-P) | 3 days
  The Numerical Rating Scale-Pain (NRS-P) is a one-dimensional tool that uses 11 numbers, ranging from 0 to 10, to assess pain intensity. The patient selects the number that most accurately reflects the severity of their pain, with 0 representing "no pain" and 10 indicating "the worst (unbearable) pain". The NRS-P is widely recognized as an effective method for measuring pain intensity, and it is generally considered more valid and reliable than other pain assessment scales.

SECONDARY OUTCOMES:
Surgical Fear Questionnaire | 3 days
  Surgical Fear Questionnaire was developed by Theunissen et al. in 2014 to determine the level of fear of short- and long-term consequences of surgery in patients who will undergo elective surgery. The scale is an 11-point Likert scale with 8 items, each scored from 0 to 10, where 0 represents "I am not scared at all" and 10 represents "I am very scared." It is divided into two sub-dimensions, each containing four items, reflecting different sources of fear. Items 1-4 assess the fear of short-term consequences of surgery, while items 5-8 focus on the fear of long-term consequences.
Safety Feeling Scale | 3 days
  Safety Feeling Scale, developed by Dabaghi et al. in 2023, is designed to assess the sense of security among hospitalized adult patients. It includes four sub-dimensions: effective care (5 items), trust in the healthcare team (3 items), emotional enrichment (2 items), and hygienic facilities (2 items), totaling 12 items. The scale uses a five-point Likert scale for responses:
  1. = Strongly disagree
  2. = Disagree
  3. = Undecided
  4. = Agree
  5. = Strongly agree Raw scale scores range from 12 to 60, with higher scores indicating a stronger sense of safety experienced by the patient in the hospital.

CONTACTS AND LOCATIONS:
Overall Officials: Yeliz CIGERCI, Assoc.Prof., Principal Investigator — Afyonkarahisar Health Sciences University
Locations (1):
- Afyonkarahisar Health Sciences University Hospital,, Afyonkarahisar, Turkey (Türkiye)